CLINICAL TRIAL: NCT04841486
Title: First Trimester of Pregnancy: Impact of a History of Miscarriage on Women's Stress
Acronym: Stress-FC
Status: Completed | Type: Observational
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-001-Stress-FC
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy
Keywords: pregnancy; women's stress; history of spontaneous termination of pregnancy
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "with history of spontaneous termination of pregnancy" group: pregnant women in the first trimester of pregnancy with history of spontaneous termination of pregnancy
  Interventions: Other: Data collection
- "without history of spontaneous termination of pregnancy" group: pregnant women in the first trimester of pregnancy without history of spontaneous termination of pregnancy
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — evaluation of women's stress

SUMMARY:
Miscarriage is the spontaneous termination of pregnancy before 22 weeks of amenorrhea. The most frequent complication of pregnancy, it represents 10 to 25% of pregnancies and affects one in four women.

Miscarriage is considered by medical personnel to be common and trivial. however, for women, it is very often a traumatic event, a source of worry for futures pregnancies.

DETAILED DESCRIPTION:
The aim of the study is to evaluate association between history of spontaneous termination of pregnancy and women's stress during the first trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* female
* pregnant (positive plasma HCG)
* in the first trimester of pregnancy
* aged 18 years old and more
* agreeing to participate in the study

Exclusion Criteria:

- less than 18 years old

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-09-11 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Women's stress | Day 0
  Women's stress evaluated using Antenatal Perceived Stress Inventory (APSI). APSI includes 12 items on medico-obstetric risks and baby's health (4 items), psychosocial changes related to pregnancy (3 items) and childbirth projections (5 items). Each item is coded from 1 to 5 points: not at all stressed, a little stressed, moderately stressed, very stressed and enormously stressed. The overall score ranges from 12 to 60 points.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra CARRAU-TRUILLET, MD, Principal Investigator — Université de Reims Champagne-Ardenne - CHU de Reims
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France